CLINICAL TRIAL: NCT02353819
Title: Phase I Clinical Trial of Stereotactic Ablative Radiotherapy (SABR) of Pelvis and Prostate Targets for Patients With High Risk Prostate Cancer
Brief Title: Stereotactic Ablative Radiotherapy (SABR) of Pelvis and Prostate Targets For High Risk Prostate Cancer
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Collaborators: National Institute for Biomedical Imaging and Bioengineering (NIBIB) (NIH)
Responsible Party: Principal Investigator, Raquibul Hannan, MD, University of Texas Southwestern Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STU 062014-027; 1R01EB027898-01 (NIH)
Record Dates: First submitted 2015-01-16; First posted 2015-02-03 (Estimated); Last update posted 2025-02-21 (Actual); Status verified 2025-02

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Stereotactic Ablative Radiotherapy (Experimental): Stereotactic Ablative Radiotherapy (SABR)
  Interventions: Radiation: Stereotactic Ablative Radiotherapy

INTERVENTIONS:
Radiation: Stereotactic Ablative Radiotherapy — SABR x5 fractions CBCT based image-guidance prior to each fraction: localize based on prostate/seeds positions SCORE system
  Other Names: SABR

SUMMARY:
Since high risk prostate cancer requires higher radiation, this study is being done to determine the maximum tolerated dose of radiation to the prostate and pelvic regions. Also to determine the feasibility and safety of each treatment fraction by using cone-beam Computed Tomography(CT) information and high speed Graphics Processing Unit based computation treatment planning systems. We also plan to determine the safety of treatment to the prostate. Health-related quality of life will be measured as part of current clinical practice.

* Determine the maximum tolerated dose (MTD) or to safely escalate dose to the pelvic nodal using 90 day acute toxicity endpoint
* Determine feasibility and safety of adaptive real time re-planning of the pelvic nodal region at each treatment fraction by using cone-beam CT (CBCT) information and high speed GPU based computation treatment planning systems
* Determine the safety and tolerability of 9.5 Gy per fraction in five fractions (47.5 Gy total dose) to the prostate
* Determine the feasibility and safety of temporal enhanced ultrasound for prostate lesion tracking during radiation therapy
* To follow tumor related outcomes (i.e. PSA control, progression-free survival (PFS), distant metastasis (DM) free survival, and overall survival (OS)
* Health-related quality of life (HRQOL) will be measured as part of current clinical practice Patients in each dose cohort will all be treated as a single group for dose escalation. There will be two levels of dose escalation-to prostate lesions and to pelvic lymph node region. Prostate/SV PTV will be treated at a fixed dose of 9.5 Gy per fraction for 5 fractions (47.5 Gy) based on our previous phase I/II study experiences. The starting dose for the dose escalation to the pelvic region PTV will be 4.5 Gy per fraction for 5 fractions (total dose= 22.5 Gy). Subsequent cohorts of patients will receive an additional 0.5 Gy per treatment (total 2.5 Gy per escalation). The starting dose for MRI-visible prostatic lesions will be 10 Gy and subsequent cohorts will receive an additional 0.5Gy per treatment (total of 2.5Gy per escalation).

DETAILED DESCRIPTION:
Patients will be accrued in alternating dose levels. The two distinct areas of dose escalations (pelvic lymph node and prostate lesion) will take place one at a time. Minimum waiting periods will be assigned between each dose cohort to observe toxicity. The phase I portion of the study will be completed when dose limiting toxicity is reached or when a sufficiently high dose level (i.e.,5.5 Gy per fraction to a total 27.5 Gy for pelvic lymph node region and 11Gy per fraction to a total of 55Gy to the prostate lesion), is attained to consider the therapy likely to be efficacious. All patients will be treated with a total of 24 months of androgen suppression therapy (ADT). Radiation therapy will start 8-12 weeks after initiation of ADT.

No. Patients for each cohort: 7-15 Cohort 1: 9.5 Gy per fraction to prostate/SV, 10 Gy per fraction to prostate lesion, 4.5Gy per fraction to pelvic lymph node region for 5 fractions for a total of 47.5 / 50 / 22.5 Gy to Prostate+SV /Prostate lesions/Nodes Cohort 2: 9.5 Gy per fraction to prostate/SV, 10 Gy per fraction to prostate lesion, 5Gy per fraction to pelvic lymph node region for 5 fractions for a total of 47.5 / 50 / 25 Gy to Prostate+SV /Prostate lesions/Nodes Cohort 3: 9.5 Gy per fraction to prostate/SV, 10.5 Gy per fraction to prostate lesion, 5Gy per fraction to pelvic lymph node region for 5 fractions for a total of 47.5 / 52.5 / 25 Gy to Prostate+SV /Prostate lesions/Nodes Cohort 4: 9.5 Gy per fraction to prostate/SV, 10.5 Gy per fraction to prostate lesion, 5.5 Gy per fraction to pelvic lymph node region for 5 fractions for a total of 47.5 / 52.5 / 27.5 Gy to Prostate+SV /Prostate lesions/Nodes Cohort 5: 9.5 Gy per fraction to prostate/SV, 11 Gy per fraction to prostate lesion, 5.5 Gy per fraction to pelvic lymph node region for 5 fractions for a total of 47.5 / 55 / 27.5 Gy to Prostate+SV /Prostate lesions/Nodes

ELIGIBILITY:
Inclusion Criteria:

* Signed study specific informed consent form.
* Patients must have at least one of the following criteria:
* The serum PSA should be greater than or equal to 20 ng/ml OR
* Study entry PSA must not be obtained during the following time frames following prostate biopsy: (2) following initiation of ADT.
* The Gleason score should be greater than or equal to 8 OR
* Eligible patients must have appropriate staging studies identifying them as AJCC stage T3+ adenocarcinoma of the prostate gland. (MR stage T3a without other high risk factors permitted at investigator discretion
* Male Patient past their 18th birthday at time of registration.
* The patient's Zubrod performance status must be 0-2
* Women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry, and during radiation treatment.
* All patients must be willing and capable to provide informed consent to participate in the protocol
* Imaging studies can include, but is not limited to the following: ultrasound, CT of pelvis/prostate (abdomen recommended) and MRI of pelvis/prostate and (abdomen recommended)
* The ultrasound, MRI or CT based volume estimation of the patient's prostate gland should not be greater than 80 grams (Repeat measurement after hormone downsizing allowed)
* Clinically negative lymph nodes, within 90 days of study enrollment, established by imaging (pelvic/prostate (abdominal recommended) CT or MRI) OR by nodal sampling OR by dissection. Nodes > 2.0 cm should be biopsied. Patients with lymph nodes equivocal or questionable by imaging are eligible if the nodes are < 2.0cm in the short axis.
* MRI Pelvis/Prostate feasible for staging and planning
* Patients with contraindications to MRI are not eligible
* Patient deemed eligible for complete androgen blockade, and androgen deprivation therapy by treating physician (this includes consideration of baseline liver function prior to initiation of therapy, if necessary at physician's discretion). For patients not eligible for anti-testosterone therapy, hormone therapy with LHRH agonist alone will be permitted on case by case by study Principal Investigator. AS can be any LHRH agonists, LHRG antagonists or anti-androgens that are approved for androgen suppression for the treatment of prostate cancer.
* Patient does not have known allergy to polyethylene glycol hydrogel (spacer material).
* Patient deemed eligible for rectal spacer ( Space OAR) placement by treating physician.
* Histologic confirmation of diagnosis of adenocarcinoma of the prostate will be required by biopsy.

Exclusion Criteria:

* Eligible patients should not have had previous pelvic radiotherapy, chemotherapy or surgery for prostate cancer.
* There must be no plans for the patient to receive other concomitant or post treatment adjuvant antineoplastic therapy while on this protocol including surgery, cryotherapy, conventionally fractionated radiotherapy, 2nd generation anti-androgen therapy (i.e Enzalutamide, Abiraterone, etc.),or chemotherapy given as part of the treatment of prostate cancer.
* The patient should not have direct evidence of regional or distant metastases after appropriate staging studies, including no distant metastases (M0) on bone scan within 90 days of study enrollment. Equivocal bone scan findings are allowed if plain films are negative for metastasis. PET or PSMA scans can be performed instead of a bone scan.
* Patients diagnosed with invasive malignancy are not eligible (except non-melanomatous skin cancer) unless disease free for a minimum of 3 years (e.g., oral cavity).
* Patients diagnosed with severe, active co-morbidity, defined as follows are not eligible:
* Unstable angina and/or congestive heart failure requiring hospitalization within the last 6 months.
* Transmural myocardial infarction within the last 6 months.
* Acute bacterial or fungal infection requiring intravenous antibiotics at the time of registration.
* Chronic Obstructive Pulmonary Disease exacerbation or other respiratory illness requiring hospitalization or precluding study therapy within 30 days before registration.
* Hepatic insufficiency resulting in clinical jaundice and/or coagulation defects; note, however, that laboratory tests for liver function and coagulation parameters are not required for entry into this protocol.
* Acquired Immune Deficiency Syndrome (AIDS) based upon current CDC definition; note, however, that HIV testing is not required for entry into this protocol. The need to exclude patients with AIDS from this protocol is necessary because the treatments involved in this protocol may be significantly immunosuppressive. Protocol-specific requirements may also exclude immuno-compromised patients.
* Patients with history of inflammatory colitis (including Crohn's Disease and Ulcerative colitis), active lupus, and scleroderma or active collagen vascular disease are not eligible.
* Patients should not have undergone previous transurethral resection of the prostate (TURP) within 1 year.
* Patients with history of inflammatory colitis (including Crohn's Disease and Ulcerative colitis) are not eligible.
* There must be no plans for the patient to receive other concomitant or post treatment adjuvant antineoplastic therapy while on this protocol including surgery, cryotherapy, conventionally fractionated radiotherapy, 2nd generation anti-androgen therapy (i.e Enzalutamide, Abiraterone, etc.),or chemotherapy given as part of the treatment of prostate cancer.
* The patient should not have direct evidence of regional or distant metastases after appropriate staging studies, including no distant metastases (M0) on bone scan within 90 days of study enrollment. Equivocal bone scan findings are allowed if plain films are negative for metastasis. PET or PSMA scans can be performed instead of a bone scan.
* Patients diagnosed with invasive malignancy are not eligible (except non-melanomatous skin cancer) unless disease free for a minimum of 3 years (e.g., oral cavity).
* Patients diagnosed with severe, active co-morbidity, defined as follows are not eligible:
* Unstable angina and/or congestive heart failure requiring hospitalization within the last 6 months.
* Transmural myocardial infarction within the last 6 months.
* Acute bacterial or fungal infection requiring intravenous antibiotics at the time of registration.
* Chronic Obstructive Pulmonary Disease exacerbation or other respiratory illness requiring hospitalization or precluding study therapy within 30 days before registration.
* Hepatic insufficiency resulting in clinical jaundice and/or coagulation defects; note, however, that laboratory tests for liver function and coagulation parameters are not required for entry into this protocol.
* Acquired Immune Deficiency Syndrome (AIDS) based upon current CDC definition; note, however, that HIV testing is not required for entry into this protocol. The need to exclude patients with AIDS from this protocol is necessary because the treatments involved in this protocol may be significantly immunosuppressive. Protocol-specific requirements may also exclude immuno-compromised patients.
* Patients with history of inflammatory colitis (including Crohn's Disease and Ulcerative colitis), active lupus, and scleroderma or active collagen vascular disease are not eligible.
* Patients should not have undergone previous transurethral resection of the prostate (TURP) within 1 year.
* Patients with history of inflammatory colitis (including Crohn's Disease and Ulcerative colitis) are not eligible.
* Patients should not have a history of significant psychiatric illness.
* Patients may have used prior hormonal therapy, but it should be limited to no more than 9 months of therapy prior to enrollment.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2015-10 (Actual); Primary Completion 2030-01 (Estimated); Study Completion 2030-12 (Estimated)

PRIMARY OUTCOMES:
maximum tolerated dose (MTD) | 90 days
  Determine the maximum tolerated dose (MTD) or to safely escalate dose to the pelvic nodal PTV using 90 day acute toxicity endpoint

SECONDARY OUTCOMES:
Adverse events | 90 days
  Determine the safety of 9.5 Gy per fraction in five fractions (47.5 Gy total dose) to the prostate/SV PTV
PSA | 5 years
  To follow tumor response to treatment
Progression-free survival | 5 years
  To follow tumor related outcomes (progression-free survival (PFS), distant metastasis (DM) free survival)
Overall survival | 5 years
  To follow tumor related outcomes , overall survival (OS)
Health-related quality of life | 5 years
  Health-related quality of life (HRQOL) will be measured as part of current clinical practice

CONTACTS AND LOCATIONS:
Overall Officials: Raquibul Hannan, MD, Principal Investigator — University of Texas Southwestern Medical Center
Locations (1):
- University of Texas Southwestern Medical Center, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No